CLINICAL TRIAL: NCT01562821
Title: A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Trial Evaluating the Safety and Efficacy of A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Trial Evaluating the Safety and Efficacy of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in Cirrhotic Patients Scheduled to Undergo Partial Hepatectomy Due to Liver Cancer or Benign Tumours
Brief Title: Safety and Efficacy of Activated Recombinant Human Factor VII in Cirrhotic Patients Undergoing Partial Hepatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7LIVER-1313
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- High dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — An initial bolus dose of 50 mcg/kg body weight (BW) followed by 50 mcg/kg BW every second hour until completion of surgery
  Arms: Low dose
Drug: activated recombinant human factor VII — An initial bolus dose of 100 mcg/kg body weight (BW) followed by 100 mcg/kg BW every second hour until completion of surgery
  Arms: High dose
Drug: placebo — An initial placebo bolus dose followed by placebo every second hour until completion of surgery
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate the haemostatic efficacy of activated recombinant human factor VII in cirrhotic patients scheduled to undergo partial hepatectomy due to liver cancer or benign tumours.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (Child-Turcotte Score A, B, or C)
* Scheduled to undergo partial hepatectomy due to liver cancer or benign tumours

Exclusion Criteria:

* Portal vein thrombosis
* Clinically documented DVT (deep venous thrombosis)
* Clinically documented symptoms of severe cardiovascular disease and/or previous myocardial/pulmonary infarction or stroke
* Present renal insufficiency requiring dialysis

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2001-07; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
The RBC transfusion requirements

SECONDARY OUTCOMES:
Number of transfusion product units
Change in coagulation-related parameters
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- China (3):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Beijing
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- [Result] Shao YF, Yang JM, Chau GY, Sirivatanauksorn Y, Zhong SX, Erhardtsen E, Nivatvongs S, Lee PH. Safety and hemostatic effect of recombinant activated factor VII in cirrhotic patients undergoing partial hepatectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Am J Surg. 2006 Feb;191(2):245-9. doi: 10.1016/j.amjsurg.2005.10.019. PMID 16442954
- [Result] Levy JH, Fingerhut A, Brott T, Langbakke IH, Erhardtsen E, Porte RJ. Recombinant factor VIIa in patients with coagulopathy secondary to anticoagulant therapy, cirrhosis, or severe traumatic injury: review of safety profile. Transfusion. 2006 Jun;46(6):919-33. doi: 10.1111/j.1537-2995.2006.00824.x. PMID 16734808
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com